CLINICAL TRIAL: NCT00110123
Title: Intravenous Versus Intra-Arterial Fotemustine Chemotherapy in Patients With Liver Metastases From Uveal Melanoma: A Randomized Phase III Study of the EORTC Melanoma Group
Brief Title: Intravenous or Hepatic Arterial Infusion of Fotemustine in Treating Patients With Unresectable Liver Metastases From Eye Melanoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-18021; EORTC-18021; 2004-002245-12 (EudraCT Number)
Record Dates: First submitted 2005-05-03; First posted 2005-05-04 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Intraocular Melanoma; Metastatic Cancer
Keywords: liver metastases; ciliary body and choroid melanoma, medium/large size; iris melanoma; extraocular extension melanoma; recurrent intraocular melanoma; metastatic intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis | interventions — fotemustine

INTERVENTIONS:
Drug: fotemustine
Drug: isolated perfusion

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fotemustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving the drugs in different ways may kill more tumor cells. It is not yet known whether giving fotemustine as an intravenous infusion is more effective than giving it as a hepatic arterial infusion in treating liver metastases.

PURPOSE: This randomized phase III trial is studying intravenous infusion of fotemustine to see how well it works compared to hepatic arterial infusion of fotemustine in treating patients with unresectable liver metastases from eye melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with surgically incurable or unresectable liver metastases secondary to uveal melanoma treated with fotemustine administered as an intravenous infusion vs an intra-arterial hepatic perfusion.

Secondary

* Compare progression-free survival of patients treated with this drug.
* Compare the response rate in patients treated with this drug.
* Compare the duration of objective response in patients treated with this drug.
* Compare the patterns of progression in patients treated with this drug.
* Compare treatment-related toxic effects and catheter-related complications in patients treated with this drug.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to participating center, lactic dehydrogenase level (normal vs abnormal), and WHO performance status (0 vs 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fotemustine IV over 1 hour on days 1, 8, and 15 (induction course). Beginning on day 50, patients receive maintenance courses of fotemustine IV over 1 hour every 21 days in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive fotemustine by a 4-hour intra-arterial (IA) hepatic perfusion on days 1, 8, 15, and 22 (induction course). Beginning on day 57, patients receive maintenance courses of fotemustine by a 4-hour IA hepatic perfusion every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 9 weeks for survival.

PROJECTED ACCRUAL: A total of 262 patients (131 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed liver metastases secondary to uveal melanoma

  * Surgically incurable or unresectable disease
* No detectable extrahepatic metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL

Hepatic

* Bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 5 times ULN
* Alkaline phosphatase < 5 times ULN
* Gamma-glutamyltransferase < 5 times ULN
* Lactic dehydrogenase < 5 times ULN

Renal

* BUN < 1.5 times ULN
* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No uncontrolled angina pectoris
* No myocardial infarction within the past 6 months
* No uncontrolled high blood pressure
* No evolutive intracranial hypertension
* No other severe cardiac disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active gastroduodenal ulcer
* No diabetes
* No active or uncontrolled infection
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up
* No other uncontrolled severe medical condition
* No other malignancy within the past 5 years except surgically cured carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunologic or biologic therapy

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for metastatic disease
* No concurrent radiotherapy

Surgery

* Recovered from prior major surgery

Other

* No prior antineoplastic drugs for metastatic disease
* More than 4 weeks since prior investigational drugs
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2005-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Duration of survival

SECONDARY OUTCOMES:
Progression-free survival
Best response as assessed by RECIST criteria
Duration of response
Toxicity as assessed by CTCAE v3

CONTACTS AND LOCATIONS:
Overall Officials: Serge Leyvraz, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (8):
- Italy (4):
  - European Institute of Oncology, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Universita di Siena, Siena
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology - Warsaw, Warsaw, Poland
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Clatterbridge Centre for Oncology, Merseyside, England
  - Ninewells Hospital, Dundee, Scotland

REFERENCES:
- [Derived] Leyvraz S, Piperno-Neumann S, Suciu S, Baurain JF, Zdzienicki M, Testori A, Marshall E, Scheulen M, Jouary T, Negrier S, Vermorken JB, Kaempgen E, Durando X, Schadendorf D, Gurunath RK, Keilholz U. Hepatic intra-arterial versus intravenous fotemustine in patients with liver metastases from uveal melanoma (EORTC 18021): a multicentric randomized trial. Ann Oncol. 2014 Mar;25(3):742-746. doi: 10.1093/annonc/mdt585. Epub 2014 Feb 7. PMID 24510314
- [Derived] Orcurto V, Denys A, Voelter V, Schalenbourg A, Schnyder P, Zografos L, Leyvraz S, Delaloye AB, Prior JO. (18)F-fluorodeoxyglucose positron emission tomography/computed tomography and magnetic resonance imaging in patients with liver metastases from uveal melanoma: results from a pilot study. Melanoma Res. 2012 Feb;22(1):63-9. doi: 10.1097/CMR.0b013e32834d3dcb. PMID 22027909